CLINICAL TRIAL: NCT00402376
Title: Effects of Combined Ventricular Unloading and Pharmacological Therapy on Left Ventricular Metabolic Dysfunction in Heart Failure
Brief Title: Evaluation of Myocardial Improvement in Patients Supported by Ventricular Assist Device Under Optimal Pharmacological Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Service de Chirurgie Cardiaque (Unknown); Institut de Physiologie, Strasbourg, France (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3212
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Heart Failure
Keywords: End-stage heart failure; heart failure;; ventricular assist device;; statin;; heart transplantation;; myocardial function;; mitochondrial respiratory function;
MeSH Terms: conditions — Heart Failure | interventions — Pravastatin; Carvedilol; Perindopril

INTERVENTIONS:
Drug: Pravastatin, Carvedilol, Perindopril
Device: Biventricular assist device (Thoratec paracorporeal assist device)

SUMMARY:
Cardiac function may improve in patients with end-stage heart failure who receive long-term support with ventricular assist devices (VAD). Reverse left ventricular remodeling may be sufficient in some cases to allow explantation of the VAD. However, some questions continue to await definitive answers. This study is designed to assess the myocardial recovery under VAD support with optimal pharmacological therapy (high doses [group I] of statins, beta-blockers, angiotensin-converting enzyme inhibitors versus standard doses [group II]).

The study is a randomized, single-blind trial performed at the Department of Cardiac Surgery, University of Strasbourg, France. Twenty patients with end-stage heart failure who will be supported by VAD (Thoratec paracorporeal device) as a bridge to heart transplantation will be included. Reverse left ventricular remodeling and myocardial function will be studied by: echocardiography, respiratory mitochondrial function, exercise testing, cardiac hormonal function, and inflammatory response. Myocardial biopsies will be obtained at the time of VAD implantation and heart transplantation. The follow-up will be performed every 4 weeks during the VAD support period. The hypothesis of this trial is that reverse left ventricular remodeling and myocardial function will improve under optimal medical therapy especially by a high dose statin.

DETAILED DESCRIPTION:
Evaluation of Myocardial Improvement (Reverse Left Ventricular Remodeling, Mitochondrial Respiratory Function) in Patients Supported by Ventricular Assist Device Under Optimal Pharmacological Therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage heart failure refractory to medical therapy and who fulfill criteria for VAD implantation as a bridge to heart transplantation
* Age > 18

Exclusion Criteria:

* Myocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
Mitochondrial function | at implantation and explantation of VAD

SECONDARY OUTCOMES:
Inflammation: IL-6; IL-8; IL-10, IL-18, TNF-α
Exercise testing : stress echocardiography, peak oxygen consumption
Hormonal cardiac function: ANP, BNP
Ventricular remodelling: echocardiography
All those parameters will be measured in the post-operative course and every 4 weeks during all the VAD support period.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Geny, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Service de Chirurgie Cardiovasculaire - Hôpital Civil, Strasbourg
  - Service de Physiologie Clinique - Hôpital Civil, Strasbourg